CLINICAL TRIAL: NCT04900155
Title: Evaluation of Long-term Lipid-lowering Therapy on Myocardial Electrical Heterogeneity, Myocardial Deformation, Arterial Stiffness and Quality of Life in Patients With Primary STEMI/NSTEMI With Coronavirus Infection COVID-19
Brief Title: Evaluation of the Effect of Long-term Lipid-lowering Therapy in STEMI Patients With Coronavirus Infection COVID-19
Acronym: CONTRAST-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Penza State University (Other)
Responsible Party: Principal Investigator, Valentin Oleynikov, Head of Therapy Department, Penza State University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSU/T-487
Record Dates: First submitted 2021-05-09; First posted 2021-05-25 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: STEMI; Covid19; NSTEMI
Keywords: myocardial strain; arterial stiffness; myocardial electrical heterogeneity; quality of life
MeSH Terms: conditions — ST Elevation Myocardial Infarction; COVID-19; Non-ST Elevated Myocardial Infarction | interventions — Atorvastatin; liptruzet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin 80 mg (Active Comparator): Initially, hypolipidemic treatment with atorvastatin at a dose of 80 mg / day is prescribed from the first 24-96 hours of myocardial infarction in addition to standard therapy for the disease.
  Interventions: Drug: Atorvastatin 80mg
- Atorvastatin-Ezetimibe (Active Comparator): In the absence of reaching the target level of LDL-C ≤1.4 mmol / L and ≥50% of the initial level after 4-6 weeks from the onset of myocardial infarction, patients additionally receive ezetimibe at a dose of 10 mg 1 time / day.
  Interventions: Drug: Atorvastatin-Ezetimibe

INTERVENTIONS:
Drug: Atorvastatin 80mg — Initially, hypolipidemic treatment with atorvastatin at a dose of 80 mg / day is prescribed from the first 24-96 hours of myocardial infarction in addition to standard therapy for the disease.
  Other Names: Atorvastatin
  Arms: Atorvastatin 80 mg
Drug: Atorvastatin-Ezetimibe — In the absence of reaching the target level of LDL-C ≤1.4 mmol / L and ≥50% of the initial level after 4-6 weeks from the onset of myocardial infarction, patients additionally receive ezetimibe at a dose of 10 mg 1 time / day.
  Other Names: Atorvastatin
  Arms: Atorvastatin-Ezetimibe

SUMMARY:
It is planned to include 200 patients hospitalized with primary myocardial infarction with and without ST segment elevation (STEMI or NSTEMI) in combination with COVID-19 within the first 15 days from the disease onset. The total follow-up period is 96 weeks.

Hypotheses:

1. An integrated approach in assessing myocardial contractility, regulation of the heart and the structural and functional state of arteries will make it possible to more accurately assess the heart pumping function; explain the mechanisms of the relationship between left ventricular (LV) contractile function and its volumetric indices; to study the mechanisms of ventriculo-arterial coupling and the influence of autonomic regulation, the role of markers of the sudden cardiac death (late ventricular potentials, pathological turbulence of the heart rate, dispersion of the QT interval).
2. In patients who have had myocardial infarction in combination with the new coronavirus infection SARS-CoV-2 (COVID-19), long-term highly effective lipid-lowering therapy, regardless of the drugs prescribed, has an antiarrhythmic effect and has a beneficial effect on the autonomic regulation of the heart rate. Highly effective lipid-lowering therapy leads to an improvement in LV contractility and structural and functional properties of the large arteries.

Methods and variables

1. Office blood pressure
2. 12-lead ECG
3. Coronary angiography. Percutaneous coronary intervention
4. Chemistry blood test
5. 2D and 3D transthoracic echocardiography (Vivid GE 95 Healthcare (USA)
6. Multi-day 3-lead ECG monitoring with assessment of the parameters of myocardial electrical instability.
7. Ultrasound of common carotid arteries using high-frequency radio-frequency signal technology
8. Applanation tonometry (SphygmoCor, AtCor, Australia)
9. Assessment of the arterial stiffness by volume sphygmography.
10. Flow-mediated vasodilation
11. Six-minute walk test
12. Computer pulse oximetry (PulseOx 7500 (SPO medical, Israel)
13. Adherence to Treatment: Counting remaining pills and completing the Morisky-Green Questionnaire
14. Assessment of quality of life
15. Assessment of physical activity: International Questionnaire On Physical Activity - IPAQ
16. Hospital Anxiety and Depression Scale (HADS)

DETAILED DESCRIPTION:
It is planned to include 200 patients hospitalized in the cardiology department of the "Penza Regional Clinical hospital Burdenko" with a STEMI diagnosis in combination with COVID-19. Patients with STEMI and NSTEMI will be included in the study within the first 15 days from the disease onset. The total follow-up period is 96 weeks.

Primary goals:

* achieving the target level of low-density lipoprotein cholesterol (LDL-C) on the background of lipid-lowering therapy as monotherapy with atorvastatin or combined treatment with atorvastatin plus ezetimibe;
* decrease in the incidence of major coronary events - percutaneous coronary interventions (PCI) / coronary artery bypass surgery (CABG) for a new case of coronary atherosclerosis, hospitalization for unstable angina or recurrent myocardial infarction;
* reduction of the frequency of life-threatening arrhythmias and markers of the risk of sudden cardiac death according to the data of long-term ECG monitoring;
* increase in myocardial contractility by improving the deformation characteristics of the peri-infarction zone.

Secondary goals:

1. Assess the effect of long-term effective lipid-lowering therapy:

   * indicators of global and regional myocardial deformation, depending on the degree of of coronary blood flow restoration according to TIMI scale;
   * systolic and diastolic LV function in the presence of initial disturbances or the absence of negative dynamics of these indicators with normal initial values;
   * on clinical and diagnostic criteria for the development or progression of heart failure (HF);
   * on the dynamics of myocardial ischemia episodes according to the data of long-term electrocardiography (ECG) monitoring;
   * for the immediate and long-term prognosis of patients;
   * on the structural and functional properties of large arteries.
2. Assess the dynamics of biochemical parameters against the background of double and monotherapy with lipid-lowering drugs.
3. Assess the safety of treatment.
4. Assess the impact on the patient's well-being and quality of life.
5. Assess therapy compliance
6. Conduct a comparative analysis of the prognostic value of markers of myocardial electrical heterogeneity, obtained from the data of long-term and 24-hour ECG monitoring.
7. To determine the effect of markers of electrical instability and autonomic regulation of cardiac activity, obtained during long-term ECG monitoring in patients at different times after myocardial infarction, on the short-term and long-term prognosis.
8. Development of a multivariate model that takes into account the parameters of electrophysiological heterogeneity and the main indicators of the cardiovascular system condition (data of echocardiography, blood vessels ultrasound, laboratory test), which allows predicting the development of repeated cardiac events.

Methods and variables

1. Office blood pressure
2. 12-lead ECG
3. Coronary angiography. Percutaneous coronary intervention
4. Chemistry blood test The lipid profile: total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), triglycerides (TG) and low-density lipoprotein cholesterol (LDL-C), non-HDL. Alanine aminotransferase (ALT), aspartat aminotransferase (AST), creatine phosphokinase (CPK), glucose, C-reactive protein (CRP), brain natriuretic peptide (BNP), serum creatinine and glomerular filtration rate (CKD-EPI), troponin I/T, CPK-MB, ferritin, sodium, potassium, lactate, procalcitonin, D-dimer, coagulogram. Nasopharyngeal swab for SARS-CoV-2 to RNA by PCR, if necessary - additional determination of immunoglobulins to SARS-CoV-2.
5. 2D and 3D transthoracic echocardiography is performed with Vivid GE 95 Healthcare (USA). The biplane ejection fraction is determined by the Simpson method, 3D ejection fraction, EDV (end-diastolic volume), ESV (end-systolic volume) and their indexed parameters in 2D and 3D mode. Left ventricular myocardial mass index (LVMI), LA volume. Myocardial deformity is analyzed using specialized software - EchoPac Software Only (General Electric Co., 2018)
6. Multi-day 3-lead ECG monitoring with assessment of the parameters of myocardial electrical instability.
7. Ultrasound of common carotid arteries using high-frequency RF signal technology will be carried out in B-mode on the MyLab 90 device (Esaote, Italy) by the following indicators: IMT - thickness of the intima-media, loc Psys - local systolic pressure in the carotid artery, loc Pdia - local diastolic pressure, P (T1) - pressure at a local point, stiffness indices β and α, DC - coefficient transverse distensibility, CC - transverse compliance coefficient, Aix - augmentation index, AR - amplification pressure, PWV - local pulse wave velocity in the carotid artery.
8. Applanation tonometry The SphygmoCor device (AtCor Medical, Australia) includes two software. The first allows to record indicators of central aortic pressure: systolic aortic pressure - SBPao, diastolic - DBPao, pulse pressure - PPao, mean hemodynamic pressure - MBPao. The PWV (pulse wave velocity) software is used to analyze the PWV in the aorta (cfPWV).
9. Assessment of the arterial stiffness by volume sphygmography. PWV in the aorta (PWV), in elastic arteries right and left (R/L-PWV) and in muscular arteries (B-PWV), Cardio-Ankle Vascular Index - CAVI.
10. Flow-mediated vasodilation
11. 6-minute walk test
12. Computer pulse oximetry (PulseOx 7500 (SPO medical, Israel)
13. Adherence to Treatment: Counting remaining pills and completing the Morisky-Green Questionnaire
14. Assessment of quality of life: Seattle Angina Questionnaire (SAQ), Minnesota LIGE with Heart Failure Questionnaire, Clinical Status Assessment Scale (CASA), analog-visual scale.
15. Assessment of physical activity International Questionnaire On Physical Activity - IPAQ
16. Hospital Anxiety and Depression Scale (HADS)

Endpoint assessment The end point is understood as the development of repeated AMI, unstable angina pectoris, PCI for a new atherosclerotic plaque, hospitalization due to chronic heart failure (CHF) exacerbation, the development of a new case of CHF II-IV NYHA class, death.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Patients of both genders aged 30 to 70 years
3. The presence of one of the options for a combination of confirmed myocardial infarction and new coronavirus infection:

3.1. Myocardial infarction that developed within 30 days from the onset of COVID-19 - in case of mild to moderate course or within 60 days - in case of severe course.

3.2. Development of a confirmed case of COVID-19 within 30 days from the myocardial infarction onset.

4.1. Clinical manifestations of acute respiratory infection (body t> 37.5 ° C and one or more signs: cough, dry or moist sputum, shortness of breath, chest tightness, SpO2 ≤ 95%, sore throat, mild or moderate rhinorrhea, impaired or loss of smell (hyposmia or anosmia), loss of taste (dysgeusia), conjunctivitis, weakness, muscle pain, headache, vomiting, diarrhea, skin rash) in the presence of at least one of the epidemiological signs:

* returning from a foreign trip 14 days before the onset of symptoms;
* having close contacts in the last 14 days with a person under surveillance for COVID-19 who subsequently fell ill;
* having close contacts in the last 14 days with a person with a laboratory confirmed diagnosis of COVID-19;
* having professional contacts with people who have a suspected or confirmed case of COVID-19.

4.2. The presence of clinical manifestations specified in 4.1, in combination with changes in the lungs according to computed tomography data, regardless of the results of a single laboratory study for the presence of SARS-CoV-2 RNA and an epidemiological history, or if it is impossible to conduct a laboratory study for the presence of SARS-RNA CoV-2.

4.3. A positive laboratory test result for the presence of SARS-CoV-2 RNA using nucleic acid amplification methods (NAA) or SARS-CoV-2 antigen using immunochromatographic analysis, regardless of clinical manifestations.

4.4. Positive result for IgA or IgM, or IgM with IgG in patients with clinically confirmed COVID-19 infection.

Primary STEMI or NSTEMI, confirmed by a diagnostically significant increase in cardiospecific enzymes (5.1) in combination with at least one criterion of acute myocardial ischemia (item 5.2):

5.1. An increase and / or decrease of serum cardiac troponin level, which should at least once exceed the 99th percentile of the URL in patients without an initial increase of serum cardiac troponin level, or its increase> 20% with an initially increased level of cardiac troponin, if up to it remained stable (variation < 20%) or declined.

5.2. Typical anginal attack / acute ischemic changes on the ECG / the appearance of pathological Q waves on the ECG / EchoCG confirmation of the presence of new areas of the myocardium with impaired local contractility / detection of intracoronary thrombosis in coronary angiography.

Presence of type 1 myocardial infarction (6.1) or type 2 (6.2), confirmed by coronary angiography:

6.1. Atherothrombosis of an infarct-related artery with a sharp decrease in blood flow distal to the damaged atherosclerotic plaque or distal embolization with thrombotic masses / fragments of atherosclerotic plaque, followed by the development of myocardial necrosis; or intramural hematoma in a damaged atherosclerotic plaque with a rapid increase in its volume and a decrease in the lumen of the artery).

6.2. Myocardial infarction developed as a result of ischemia caused by non-thrombotic complications of coronary atherosclerosis. Pathophysiologically, such myocardial infarctions are associated with an increase in myocardial oxygen demand and / or a decrease in its delivery to the myocardium, for example, due to coronary artery embolism, spontaneous coronary artery dissection, respiratory failure, anemia, cardiac arrhythmias, arterial hypertension or hypotension, etc.

Duration of subsequent hospitalization after inclusion in the study - at least 5 days

Exclusion Criteria:

1. Hemodynamically significant stenosis of the left coronary artery> 30%.
2. Recurrent or repeated STEMI or NSTEMI.
3. Exogenous hypertriglyceridemia (type 1 hyperchylomicronemia - TC / TG <0.15).
4. Acute heart failure III-IV.
5. Individual intolerance to statins, ezetimibe, alirocumab.
6. Congenital and acquired heart defects.
7. Non-sinus rhythm, artificial pacemaker.
8. Sinoatrial and atrioventricular block of 2-3 degrees.
9. QRS complex> 100 ms.
10. Complete blockade of left or right bundle branch.
11. History of CHF III-IV class according to NYHA.
12. The presence of pronounced LV hypertrophy according to echocardiography (IVS / LVS> 14 mm).
13. Uncontrolled hypertension with SBP> 180 mm Hg. and DBP> 110 mm Hg.
14. Diabetes mellitus type 1 or type 2 requiring insulin therapy.
15. Presence of anemia at the time of screening (Hb <100 g / l)
16. Chronic kidney disease (GFR < 30 ml / min / 1.73 m2 according to the CKD-EPI formula).
17. Uncorrected thyroid dysfunction in the presence of hyper- / hypothyroidism.
18. Body mass index (BMI) ≥35 kg / m2.
19. Pregnancy, lactation.
20. Alcohol abuse, drug use.
21. Other severe concomitant diseases that exclude the possibility of participation in the study.
22. Participation in other clinical trials within the previous 2 months.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Lipid profile assessment | up to 96 weeks
  Achievement of target level of lipid profile (total cholesterol, LDL-С, HDL-C, triglycerides) during the atorvastatin therapy
Assessment of ventricular rhythm disturbances | up to 96 weeks
  The frequency of ventricular arrhythmias recorded with 24 hour ECG monitoring
Electrical instability and autonomic regulation of heart rate | up to 96 weeks
  Changes in parameters of electrical instability and autonomic regulation of heart rate recorded with 24 hour ECG monitoring
Left ventricular systolic function | up to 96 weeks
  Assessment of LV systolic function differences according to echocardiography during atorvastatin treatment
Left ventricular myocardial deformation (strain, strain rate) | up to 96 weeks
  Assessment of LV myocardial deformation (strain, strain rate) differences according to echocardiography during atorvastatin treatment
Number of Participants with major cardiovascular events | up to 96 weeks
  Number of Participants with major cardiovascular events: PCI / CABG for a new case of coronary atherosclerosis, hospitalizations for unstable angina pectoris, recurrent AMI

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Oleynikov, Principal Investigator — Penza State University
Locations (1):
- Valentin Oleynikov, Penza, Russia